CLINICAL TRIAL: NCT05717062
Title: Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of Intravenous Varespladib Followed by Oral Varespladib in Addition to Standard of Care in Subjects Bitten by Venomous Snakes
Brief Title: Broad-spectrum Rapid Antidote: Varespladib IV to Oral Trial for Snakebite (BRAVIO)
Acronym: BRAVIO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ophirex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPX-PR-03; FD-R-7839 (Other Grant/Funding Number: FDA-OOPD)
Record Dates: First submitted 2023-01-20; First posted 2023-02-08 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Snakebite; Envenoming, Snake
Keywords: Envenoming, Snakebite, varespladib; antidote; snake
MeSH Terms: conditions — Snake Bites | interventions — varespladib; varespladib methyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Varespladib Intravenous Form (IV) + Varespladib Oral tablet (LY315920) + SOC (Experimental): Participants will receive intravenous (IV) infusion of varespladib at dose of 0.45 milligrams per kilogram per hour (mg/kg/hr) for six hours. This infusion will continue until when the participant meets clinical criteria for transition to oral drug, -If criteria are met, they will be transitioned to varespladib-methyl (initial dose of 500 mg) then continued oral dosing q12 (once every 12 hours) of 250 mg for the remainder of the study period. Participants that do not meet the criteria for transitioning to the oral drug will remain on the IV infusion at 0.45 mg/kg/hr (along with SOC) and assessed twice a day until they meet criteria for transition to oral drug.
  Interventions: Drug: Varespladib intravenous form; Drug: varespladib-methyl- oral form
- Placebo Intravenous (IV) + Placebo Oral + SOC (Active Comparator): Participants will receive intravenous (IV) infusion of placebo matched to varespladib for six hours. This infusion will continue until the participant meets clinical criteria for transition to oral drug. If criteria are met, they will be transitioned to the oral placebo then continued oral dosing for the remainder of the study period. Participants that do not meet the criteria for transitioning to the oral drug will remain on the IV infusion (along with SOC) and assessed twice a day until they meet criteria for transition to oral drug.
  Interventions: Drug: Placebo intravenous form; Drug: Placebo - oral form

INTERVENTIONS:
Drug: Varespladib intravenous form — This is a lyophilized drug contained in 100 mg vials to be reconstituted in Water for Injection (WFI), followed by dilution into 0.9% Sodium Chloride Injection.
  Other Names: LY315920
  Arms: Varespladib Intravenous Form (IV) + Varespladib Oral tablet (LY315920) + SOC
Drug: varespladib-methyl- oral form — Varespladib-methyl (LY333013) is an immediate-release, oval, white, film-coated tablet at a dosage strength of 250 mg for oral administration.
  Other Names: LY333013
  Arms: Varespladib Intravenous Form (IV) + Varespladib Oral tablet (LY315920) + SOC
Drug: Placebo intravenous form — The intravenous placebo will be saline (0.9%). Blinding will be ensured by covering the bag containing the investigational product with opaque covers.
  Arms: Placebo Intravenous (IV) + Placebo Oral + SOC
Drug: Placebo - oral form — Oral placebo is supplied as a white film-coated oval tablet to match the appearance of the LY333013 250 mg tablet and contains a subset of the excipients present in the active tablet formulation: lactose monohydrate, microcrystalline cellulose, and magnesium stearate
  Arms: Placebo Intravenous (IV) + Placebo Oral + SOC

SUMMARY:
This is a multicenter,randomized,double-blind, placebo-controlled, phase 2 study designed to evaluate the safety, tolerability and efficacy of a continuous rate infusion (CRI) of IV varespladib followed by transition to the oral dosage form, varespladib-methyl, concurrently with SOC, in participants bitten by venomous snakes.

Note: Funding Source - FDA-OOPD

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, phase 2 study designed to evaluate the safety, tolerability and efficacy of intravenous varespladib followed by oral varespladib, concurrently with standard of care (SOC), in participants bitten by venomous snakes.

Approximately 140 male and female eligible participants will be enrolled and randomized to receive active varespladib or placebo (in addition to SOC)

Randomization will be stratified by the presence or absence of neurotoxicity (SSS nervous system subscore of 0-1 or ≥ 2) at Baseline, and by receipt of antivenom prior to screening, resulting in 4 strata in total.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Is a male or female ≥ 18 years of age with venomous snakebite.
2. Patients must have known or suspected venomous snakebite. In India, enrollment will be restricted to patients bitten by suspected or confirmed Russell's viper (Daboia russelii) or krait (Bungarus spp.) In the U.S., any snakebite that meets all other criteria may be eligible.
3. Participants must meet one of two categories of inclusion criteria:

   1. Category 1: The participant is enrolled within 5 hours of venomous snakebite or symptom onset with an SSS score of ≥2 in one system and ≥1 in another system (2+1).

      OR
   2. Category 2: The participant has a suspected or confirmed bite from an elapid and is enrolled within 10 hours of bite or symptom onset with moderate to severe cranial nerve or skeletal muscle weakness.
4. Is willing (or legally authorized representative is willing) to provide informed consent prior to initiation of any study procedures.

EXCLUSION CRITERIA:

1. Has history of or is suspected to have CVA or intracranial bleeding of any kind, acute coronary syndrome, MI, or severe pulmonary hypertension.
2. Has known history of inherited bleeding or coagulation disorder.
3. Is, at Screening Visit, using the following anticoagulants: warfarin/coumadin, argatroban, bilvalirudin, lepirudin, apixaban, dabigatran, clopidogrel, prasugrel, ticlodipine or another anticoagulant agent not specifically listed, or has used heparin, enoxaparin, fondaparinux, or other low molecular weight heparin or any antiarrhythmic drugs within 14 days prior to treatment.
4. Has a history of chronic liver disease such as chronic active viral hepatitis, alcohol- related liver disease, non-alcoholic steatohepatitis, non-alcoholic fatty liver disease, hemochromatosis, primary biliary cirrhosis, primary sclerosing cholangitis, autoimmune hepatitis.
5. Reports or has known pre-existing renal impairment or chronic kidney disease.
6. Has a known allergy or significant adverse reaction to varespladib or varespladib-methyl.
7. Is considered by the Investigator to be unable to comply with protocol requirements due to geographic considerations, psychiatric disorders, or other compliance concerns.
8. Is pregnant, has a positive serum human chorionic gonadotropin (hCG) pregnancy test or not willing to use a highly effective method of contraception for 14 days after initial treatment, or is breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
For subjects bitten by vipers: Area Under the Curve (AUC) of an abbreviated Snakebite Severity Score | Baseline to Day 14
  For subjects bitten by vipers: Area Under the Curve (AUC) of an abbreviated Snakebite Severity Score (SSS) composed of local wound, hematologic, and neurologic subscores from Baseline (pre-dosing) to Day 14.
  The independent p-values from subjects bitten by elapids and subjects bitten by vipers will be analyzed using Fisher's combined probability test to obtain a single global p-value for testing the primary endpoint.
  The Snakebite Severity Scale is a tool used to measure the severity of envenoming, a higher score indicates worse symptoms.
For subjects bitten by elapids: Time to complete head-lift recovery defined by a 5-second head-lift of 5 seconds. | Baseline to Day 14
  The independent p-values from subjects bitten by elapids and subjects bitten by vipers will be analyzed using Fisher's combined probability test to obtain a single global p-value for testing the primary endpoint.

SECONDARY OUTCOMES:
Area under the curve of the composite outcome of pulmonary, cardiovascular, local wound, hematologic, renal, and nervous system sections of the SSS from Baseline to Day 7, among patients randomized within 5 hours from bite. | Baseline to Day 7
  The SSS is a tool developed to measure the severity of snakebite envenoming. Each category is graded from 0 to 3 or 4 (depending on the body category) and a higher score indicates worse signs or symptoms.
Patient Specific Functional Scale (PSFS) score at Day 3 and Day 7. | Day 3 and Day 7
  Patient Specific Functional Scale (PSFS) is a brief, interview-format questionnaire that is used to assess functional disability and any changes in performance of activities. The patient provides 3 activities. The patient then provides a rating for each item on an 11-item ordinal scale, where 0 is "unable to perform activity" and 10 is "able to perform activity at the same level as before injury or problem." The range of possible single activity scores is 0 to 10 and the range of possible total score is 0 to 10 (0 is unable to perform and 10 is perform as before injury/illness).
Complete Snakebite Severity Scale Score (SSS) recovery, from baseline to Day 28. | Baseline through Day 28
  Complete snakebite severity score (SSS) recovery, defined as a composite score of 0 for the pulmonary, cardiovascular, local wound, hematologic, renal, and nervous system sections of the SSS at Day 28. The SSS is a tool developed to measure the severity of snakebite envenoming. Each category is graded from 0 to 3 or 4 (depending on the body category) and a higher score indicates worse signs or symptoms.
Total Antivenom Requirement, measured in number of vials of antivenom administered to the subject, from baseline (pre-dosing) through Day 28 | Baseline through Day 28
Duration of Hospitalization from baseline (pre-dosing) through Day 28 | Baseline through Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Platts-Mills, MD, MSc, Principal Investigator — Ophirex, Inc.
Locations (10):
- United States (10):
  - Banner University Medical Center - Phoenix, Phoenix, Arizona
  - Arizona Poison & Drug Information Center, Tucson, Arizona
  - Desert Regional Medical Center, Palm Springs, California
  - Antelope Valley Medical Center, Rosamond, California
  - UF Health Shands Hospital, Gainesville, Florida
  - University of South Florida/Tampa General Hospital, Tampa, Florida
  - Emergency Medicine, University of Kentucky, Lexington, Kentucky
  - Duke University Medical Center, Durham, North Carolina
  - Texas Tech University Health Sciences Center El Paso, El Paso, Texas
  - UT Health San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No